CLINICAL TRIAL: NCT01785342
Title: Detection of Early Lung Cancer Among Military Personnel Study 1 (DECAMP-1): Diagnosis and Surveillance of Indeterminate Pulmonary Nodules
Brief Title: DECAMP-1: Diagnosis and Surveillance of Indeterminate Pulmonary Nodules
Acronym: DECAMP-1
Status: Completed | Type: Observational
Sponsor: Boston University (Other)
Collaborators: American College of Radiology Imaging Network (Network); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: H-31755; U01CA196408 (NIH)
Record Dates: First submitted 2013-02-05; First posted 2013-02-07 (Estimated); Last update posted 2022-03-15 (Actual); Status verified 2022-02

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Blood Specimen Collection; Urination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Urine, Sputum, Nasal brushing, Buccal scraping, Bronchial Biopsy, Bronchial brushing, lung tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Indeterminate Pulmonary Nodule: The goal will be accomplished by recruiting 500 smokers with indeterminate pulmonary nodules (0.7cm - 3.0cm) on chest CT who will undergo fiberoptic bronchoscopy and will be followed for 2 years until a final diagnosis is made. Biosample and imaging collection will be done.
  Interventions: Other: Biosample and Imaging Collection

INTERVENTIONS:
Other: Biosample and Imaging Collection — Collection of listed biosamples and CT imaging.
  Other Names: Blood,; Urine,; Buccal Scraping,; Nasal,; Bronchial Brushing,; Bronchial Biopsy,; Lung Tissue,; Sputum,; CT Imaging of Chest

SUMMARY:
The goal is to improve the efficiency of the diagnostic follow-up of patients with indeterminate pulmonary nodules by determining whether biomarkers for lung cancer diagnosis that are measured in minimally invasive biospecimens are able to distinguish malignant from benign pulmonary nodules that are incidentally detected in high-risk smokers.

DETAILED DESCRIPTION:
The Detection of Early lung Cancer Among Military Personnel (DECAMP) consortium is a multidisciplinary and translational research program that includes 7 Veterans Administration Hospitals (VAH), the 4 designated Military Treatment Facilities (MTF) and 4 academic hospitals as clinical study sites, several molecular biomarker laboratories, along with Biostatics, Bioinformatics, Pathology and Biorepository cores. The DECAMP Coordinating Center will facilitate rapid selection, design and execution of clinical studies within this multi-institutional consortium. The goal will be accomplished by recruiting 500 smokers with indeterminate pulmonary nodules (0.7cm - 3.0cm) on chest CT who will undergo fiberoptic bronchoscopy and will be followed for 2 years until a final diagnosis is made. The diagnostic performance of four previously established lung cancer biomarkers in this cohort will be validated; 1) a gene-expression biomarker measured in bronchial airway brushings; 2) a proteomic signatures measured in bronchial airway biopsies; 3) a proteomic signature measured in serum; and 4) a signature of serum cytokines. The added value of the molecular markers to clinical and imaging markers routinely used in the diagnostic work up of these patients and develop an integrated model (i.e. clinical, imaging & molecular markers) that results in the most robust diagnostic predictor will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 45 years of age or older;
* Initial diagnosis of indeterminate pulmonary nodule (0.7-3.0 cm);
* Smoking status: Current or former smoker with ≥ 20 pack years (pack years = number of packs per day X number of years smoked)
* Willing to undergo fiberoptic bronchoscopy;
* Able to tolerate all biospecimen collection as required by protocol;
* Able to comply with standard of care follow up visits including clinical exams, diagnostic work-ups, and imaging for a minimum of two years;
* Able to fill out Patient Lung History questionnaire;
* Willing and able to provide a written informed consent.

Exclusion Criteria:

* History or previous diagnosis of lung cancer;
* Diagnosis of pure ground glass opacities on chest CT;
* Contraindications to nasal brushing or fiberoptic bronchoscopy including ulcerative nasal disease, hemodynamic instability, severe obstructive airway disease, unstable cardiac or pulmonary disease; inability to protect airway or altered level of consciousness;
* Allergies to any local anesthetic that may be used to obtain biosamples in the study.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Military personnel
Sampling Method: Non-Probability Sample
Enrollment: 489 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Lung Cancer | 2 years
  Subjects will be identified as Lung Cancer or no Lung Cancer (through diagnosis) within the 2 year followup period.

CONTACTS AND LOCATIONS:
Overall Officials: Ehab Billatos, MD, Principal Investigator — Boston University; Deni Aberle, MD, Principal Investigator — University of California, Los Angeles
Locations (15):
- United States (15):
  - Regents of the University of California LA (Los Angeles VA Healthcare System), Los Angeles, California
  - University of California Los Angeles Medical Center, Los Angeles, California
  - Naval Medical Center San Diego, San Diego, California
  - Denver Research Institute, Denver, Colorado
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Boston University Medical Center, Boston, Massachusetts
  - Boston VA Research Institute, Inc, Boston, Massachusetts
  - Health Research Inc. Roswell Park Division, Buffalo, New York
  - Trustees of University of Pennsylvania (Philadelphia VA Medical Center), Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Veterans Research Foundation of Pittsburgh, Pittsburgh, Pennsylvania
  - Middle Tennessee Research Institute (Vanderbilt University), Nashville, Tennessee
  - Dallas VA Research Corporation, Dallas, Texas
  - San Antonio Military Medical Center, San Antonio, Texas
  - Naval Medical Center Portsmouth, Portsmouth, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kinsey CM, Billatos E, Mori V, Tonelli B, Cole BF, Duan F, Marques H, de la Bruere I, Onieva J, San Jose Estepar R, Cleveland A, Idelkope D, Stevenson C, Bates JHT, Aberle D, Spira A, Washko G, San Jose Estepar R. A simple assessment of lung nodule location for reduction in unnecessary invasive procedures. J Thorac Dis. 2021 Jul;13(7):4207-4216. doi: 10.21037/jtd-20-3093. PMID 34422349
- [Derived] Billatos E, Ash SY, Duan F, Xu K, Romanoff J, Marques H, Moses E, Han MK, Regan EA, Bowler RP, Mason SE, Doyle TJ, San Jose Estepar R, Rosas IO, Ross JC, Xiao X, Liu H, Liu G, Sukumar G, Wilkerson M, Dalgard C, Stevenson C, Whitney D, Aberle D, Spira A, San Jose Estepar R, Lenburg ME, Washko GR; DECAMP and COPDGene Investigators. Distinguishing Smoking-Related Lung Disease Phenotypes Via Imaging and Molecular Features. Chest. 2021 Feb;159(2):549-563. doi: 10.1016/j.chest.2020.08.2115. Epub 2020 Sep 16. PMID 32946850
- [Derived] Billatos E, Duan F, Moses E, Marques H, Mahon I, Dymond L, Apgar C, Aberle D, Washko G, Spira A; DECAMP investigators. Detection of early lung cancer among military personnel (DECAMP) consortium: study protocols. BMC Pulm Med. 2019 Mar 7;19(1):59. doi: 10.1186/s12890-019-0825-7. PMID 30845938